CLINICAL TRIAL: NCT00156390
Title: Predictors of Response to Biventricular Pacing in Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samir Saba (Other)
Responsible Party: Sponsor-Investigator, Samir Saba, Director, Cardiac Electrophysiology, UPMC, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0504006; 0504006
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2014-11-24 (Estimated); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Heart Failure, Wide QRS Complex
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): echo-guided LV lead placement
  Interventions: Device: echo-guided left ventricular lead placement
- 2 (Other): LV lead placement as per standard of care (without echo-guidance)
  Interventions: Other: LV lead placement as per standard of care (without echo guidance)

INTERVENTIONS:
Device: echo-guided left ventricular lead placement — placement of the LV lead of the biventricular pacing device under echocardiographic guidance
  Arms: 1
Other: LV lead placement as per standard of care (without echo guidance)
  Arms: 2

SUMMARY:
Heart Failure (HF) is a disease of epidemic proportion in the U.S. affecting over 5 million individuals. It is estimated that in the next year nearly 400,000 new cases will be diagnosed, 1 million individuals will be hospitalized and 300,000 deaths will occur because of HF. Approximately half of the deaths will be attributed to worsening pump function while the remainder will be attributable to sudden cardiac death.

Biventricular (BIV) pacing has recently emerged as an exciting new treatment of advanced HF with dramatic benefits to some patients. Current candidates include those with ventricular conduction abnormalities and reduced ejection fraction who continue to suffer from severe HF symptoms despite optimal pharmacological therapy. Recent clinical trials have demonstrated that BIV pacing improves myocardial function, functional capacity, quality of life, as well as reduces the incidence of hospitalization and even prolongs life. Despite all this, about one third of patients with HF do not benefit from BIV pacing, the so-called 'non-responders'. Our group and others have shown that there are direct genetic effects of BiV pacing in an animal model, however, there are gaps in existing knowledge about the effects of left ventricular (LV) pacing site or genetic influences on the degree of response to this novel therapy.

This proposal aims at identifying predictors of benefit from Biventricular (BIV) pacing with the goal of optimizing the degree of benefit and increasing the proportion of patients who respond to this therapy. Patients who fulfill current indications for BIV pacing will undergo and echocardiography (echo) with regional tissue Doppler analysis and cardiac imaging consisting of a myocardial perfusion imaging(EGC rest gated Spect scan using Sestamibi) prior to implantation of a BIV pacing device. They will then be randomly assigned to empiric versus echo and Spect scan-guided LV lead positioning. In this latter group, optimal LV pacing site will be defined as the site of latest peak tissue velocity by tissue Doppler echo and Spect scan testing. In the empiric group, the LV lead position will be chosen by the masked operator based on the coronary sinus venous anatomy, on electrocardiographic (ECG) criteria, or other as per standard of care. Blood would be collected from all patients at the time of the procedure for analysis of genetic polymorphisms.

DETAILED DESCRIPTION:
1. To test the hypothesis that the number, size, location, and severity of myocardial perfusion defects and scar distribution dictate the pattern of LV dyssynchrony by tissue Doppler echocardiography and speckle tracking. An extensive body of literature exists describing the predictors of response to BIV pacing in HF patients. Our group and others have established a clear association between the presence of mechanical cardiac dyssynchrony and the response to BIV pacing. Also, our group and others have examined the effect defects on myocardial perfusion imaging (MIBI) scan on response to BIV pacing. What remains unclear is the relationship between the number, size, distribution, and severity of these perfusion defects and the pattern of dyssynchrony by echo. It seems plausible that the distribution of scar and/or perfusion abnormalities dictates the pattern of mechanical delay and the relative timing of contraction of the various parts of the LV. Approach: In this first phase of the proposal, we will utilize some of the techniques that are available to our group to correlate the patterns of perfusion defects with the patterns of mechanical dyssynchrony. For that purpose, patients with clinical indications for BIV pacing will undergo nuclear perfusion imaging at rest as well as echocardiographic (echo) imaging with tissue Doppler assessment and speckle tracking. The site of latest mechanical activation and pattern of mechanical contraction will then be compared to the sites of scar and/or perfusion defects on the resting MIBI scan. Anticipated Results: The purpose of this first phase of the proposal would be to identify if the dyssynchrony pattern is a downstream manifestation of the myocardial injury scheme and therefore, if it can be predicted based on the number, size, severity, and distribution of the perfusion abnormalities.
2. To test the hypothesis that LV lead positioning away from dense scars as determined by resting nuclear perfusion imaging and close to the site of latest LV mechanical activation translates into improved response after BIV pacing. Our group and others have demonstrated improved acute hemodynamics and long term response to BIV pacing if the LV lead position was concordant with the site of latest mechanical activation of the LV. Also, our group and others have shown that an LV pacing lead positioned at the site of a scar or in the vicinity of a high scar density area is associated with little echocardiographic and clinical response after BIV pacing. To date, standard clinical practice continues to consist of placing the LV lead tip in the most lateral and posterior position. Maintaining this approach in all cardiomyopathy patients regardless of the nature of the myocardial insult or the sites of scaring may not be optimal and may account for the lack of response to BIV therapy in a significant number of patients. The primary objective of this specific aim is to demonstrate that MIBI/echo-guided LV lead placement is superior to standard lead placement and that patients who are randomized to the MIBI/echo-guided arm will exhibit greater improvement in the symptoms of HF and greater improvement of LV function at the 6-month interval compared to patients receiving standard LV lead placement. Approach: Heart failure patients (n=210) enrolled in this study will be randomly assigned in a 2:1 fashion to one of two study arms:

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years Heart Failure Ejection fraction<35% QRS complex>120 ms

Exclusion Criteria:

* pregnant unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Saba S, Marek J, Schwartzman D, Jain S, Adelstein E, White P, Oyenuga OA, Onishi T, Soman P, Gorcsan J 3rd. Echocardiography-guided left ventricular lead placement for cardiac resynchronization therapy: results of the Speckle Tracking Assisted Resynchronization Therapy for Electrode Region trial. Circ Heart Fail. 2013 May;6(3):427-34. doi: 10.1161/CIRCHEARTFAILURE.112.000078. Epub 2013 Mar 8. PMID 23476053
- See also: Related Info — http://circheartfailure.ahajournals.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Echo-guided LV Lead Placement: echo-guided LV lead placement
  echo-guided left ventricular lead placement: placement of the LV lead of the biventricular pacing device under echocardiographic guidance
- LV Lead Placement as Per Standard of Care (Without Echo-guida: LV lead placement as per standard of care (without echo-guidance)
  placement of the LV lead of the biventricular pacing device without echocardiographic guidance
Period: Overall Study
Arm/Group | Echo-guided LV Lead Placement | LV Lead Placement as Per Standard of Care (Without Echo-guida
Started | 110 | 77
Completed | 96 | 69
Not Completed | 14 | 8

BASELINE CHARACTERISTICS:
Groups:
- LV Lead Placement as Per Standard of Care (Without Echo-guidan: LV lead placement as per standard of care (without echo-guidance)
  placement of the LV lead of the biventricular pacing device without echocardiographic guidance
- Total: Total of all reporting groups
Arm/Group | Echo-guided LV Lead Placement | LV Lead Placement as Per Standard of Care (Without Echo-guidan | Total
Number analyzed (Participants) | 110 | 77 | 187
Age, Continuous [Mean (Full Range); unit: years] | 66 [55 to 77] | 67 [54 to 80] | 66.5 [54 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 17 | 50
  Male | 77 | 60 | 137
Region of Enrollment [Number; unit: participants]
  United States | 110 | 77 | 187

OUTCOME MEASURES:

1. Primary Outcome: Minnesota For Living With Heart Failure Questionnaire
Description: Quality of Life Questionnaire List of 21 Questions; each question has a Scale 0-5 with 0 = "no" heart failure did not prevent one from living as they want and 5= "yes"heart failure prevented one very much from living as they want. Overall scores between 0-105, with 105 being the worse quality of life.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Echo-guided LV Lead Placement | LV Lead Placement as Per Standard of Care (Without Echo-guidan
Number analyzed (Participants) | 96 | 69
units on a scale | 31 (26) | 24 (20)

2. Secondary Outcome: Echocardiographic Changes
Description: These parameters compared the echocardiographic measures at baseline prior to device implantations to those obtained 6 to 12 months after device implantation. Data for ESV and EF are presented as percent relative change (standard deviation)
Time Frame: 1 year
Population: Echo Results. The numbers in the outcome measure data table represent the patients who had both baseline and follow-up echo data. Patients who died or were lost to follow-up before having their follow-up echocardiogram are not included in this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Echo-guided LV Lead Placement | LV Lead Placement as Per Standard of Care (Without Echo-guida
Number analyzed (Participants) | 87 | 62
percent change
  Relative change in ESV (standard deviation) | -30 (29) | -20 (25)
  Relative change in EF (standard deviation) | 12 (11) | 9 (10)

ADVERSE EVENTS:
Arm/Group | Echo-guided LV Lead Placement | LV Lead Placement as Per Standard of Care (Without Echo-guidan
Serious Adverse Events (participants affected / at risk) | 31/110 | 36/77
Other Adverse Events (participants affected / at risk) | 8/110 | 7/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Echo-guided LV Lead Placement (N=110) | LV Lead Placement as Per Standard of Care (Without Echo-guidan (N=77)
Death (Cardiac disorders) | 15 | 15
Heart Failure Hospitalization (Cardiac disorders) | 16 | 21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Echo-guided LV Lead Placement (N=110) | LV Lead Placement as Per Standard of Care (Without Echo-guidan (N=77)
Device infection (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
pneumothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LV lead dislodgement (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Atrial Lead Dislodgement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
coronary sinus staining during venography (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
diaphragmatic stimulation from LV pacing requiring device reprogramming (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes